CLINICAL TRIAL: NCT07254377
Title: START: Design and Validation of Innovative Strategies Based on Dual-Task Approach for Neuro- Rehabilitation Technologically-supported in People With Chronic Neuro-inflammatory Disease
Brief Title: Design and Validation of Innovative Strategies Based on Dual-Task Approach
Acronym: START
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: Vito Fazzi Hospital (Unknown); ASL Frosinone (Unknown); Azienda Ospedaliera San Giovanni di Dio Ruggi d'Aragona (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNRR-MCNT2-2023-12378271
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Multiple Sclerosis; Parkinson Disease; Dual Task Exercises; Long COVID
Keywords: dual task; cognitive motor integration; neurological disease; validation
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Parkinson Disease; Post-Acute COVID-19 Syndrome; Nervous System Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Dual Task training) (Experimental): The dual-task rehabilitation program includes a series of progressively complex activities targeting upper-limb function, balance, motor imagery, and gait.
  Interventions: Other: Dual Task exercise
- Control Group (conventional motor exercises) (Active Comparator): Patients in the control group will perform stationary cycling (or an equivalent low-resistance aerobic activity) instead of the dual-task training.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Dual Task exercise — Upper-limb sessions employ Virtual Art Therapy, during which the seated patient performs virtual painting tasks that simultaneously stimulate motor control and cognitive engagement. Balance training initially requires the patient to stand still with eyes closed-sometimes on unstable surfaces-while performing serial subtraction tasks, followed in later sessions by the Fukuda stepping test combined with the identification of male or female voices presented in congruent or incongruent sequences. Motor imagery sessions involve imagining the number of steps and time needed to reach a cone placed at varying distances before executing the actual movement. Gait training, conducted overground or on a treadmill, integrates various cognitive challenges: generating lists from semantic categories, recognizing objects or colors in the environment, repeating short word sequences for memory engagement, performing serial subtraction while walking, responding to directional auditory stimuli.
  Arms: Experimental Group (Dual Task training)
Other: Physical therapy — Conventional exercises for upper and lower limbs motor rehabilitatiion
  Arms: Control Group (conventional motor exercises)

SUMMARY:
People affected by Stroke, Multiple Sclerosis (MS), and Parkinson's disease (PD) share severe and complex disabilities. Widespread neuro-inflammatory processes represent an important pathogenetic component in all three conditions. The potential overlap with neurological complications of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection has further contributed to the worsening of functional impairment. Since pharmacological therapies have limited or negligible effects in these disorders, neurorehabilitation plays a crucial role in restoring and maintaining adequate functional abilities. In this context, dual-task strategies have attracted growing interest, but their effectiveness has not been adequately assessed in the above neurological conditions-and not at all in individuals with long-term sequelae of SARS-CoV-2 infection.

Based on these premises, the objectives of this research project are:

* to design rehabilitation strategies using the dual-task approach in its various forms (dual motor task, dual cognitive task, and combined motor-cognitive task) and to conduct feasibility tests in small groups of individuals affected by stroke, MS, PD, or long-term Coronavirus Disease 2019 (COVID-19) sequelae;
* to apply the strategies found to be effective in larger trials involving participants with stroke, MS, or PD, with or without a history of SARS-CoV-2 infection;
* to compare the outcomes of dual-task strategies with those obtained through conventional rehabilitation approaches.

The activities planned within the project will be distributed among the four participating operating units (OUs). OU1 (Santa Lucia Foundation) will be responsible for:

1. designing and validating dual-task rehabilitation strategies covering the three possible combinations of motor and cognitive activities (dual motor task, dual cognitive task, and combined motor-cognitive task);
2. assessing the feasibility of these strategies through a pilot study involving small groups of individuals with the aforementioned neurological conditions, including those with long-term outcomes of SARS-CoV-2 infection, and selecting the most suitable approaches.

All four OUs will participate in the selection and enrollment of subjects for the trial phase.

OUs 1, 3, and 4 (Collaborators to the project) will conduct the activities planned for the experimental trial, including:

1. baseline assessment of enrolled participants using validated instruments to measure various motor and cognitive functions;
2. implementation of rehabilitation strategies based on the dual-task approach, making use of newly emerging technological devices;
3. follow-up assessments at the end of the treatment period and again three months later.

Assessments will focus on motor functions such as gait and balance, cognitive functions, mood, the occurrence of domestic accidents, and the measurement of circulating biomarkers of neuroinflammation and neurodegeneration.

Data collected throughout the different phases of the study will be compiled into a single database, and statistical analyses will be performed by researchers from OU1.

The interpretation of results will be carried out collaboratively by members of all OUs, and findings will be disseminated through participation in conferences and congresses, as well as through publications in peer-reviewed international indexed journals.

DETAILED DESCRIPTION:
Summary Description

Neurological diseases such as Stroke Outcomes (SO), Multiple Sclerosis (MS), and Parkinson's disease (PD) cause complex and severe disabilities involving motor, cognitive, and autonomic domains. Widespread neuroinflammation contributes to progressive tissue damage in all three conditions. SARS-CoV-2 infection can further exacerbate neurological deficits through inflammatory mechanisms, and its long-term effects may aggravate pre-existing motor and cognitive impairments. Pharmacological therapies for these diseases-and for post-COVID neurological sequelae-offer limited benefit; therefore, neurorehabilitation represents a crucial therapeutic resource.

Dual-task approaches, which simultaneously target cognitive and motor functions, have gained increasing interest because they better reflect daily life demands, align with embodied cognition theories, and allow concurrent intervention on multiple deficit domains. However, their efficacy has not been adequately assessed in SO, MS, and PD, and has not been investigated at all in individuals with long-term neurological consequences of SARS-CoV-2. This project aims to design and validate dual-task rehabilitation strategies in these populations and compare their outcomes with those of conventional rehabilitation.

Background and State of the Art

Individuals with SO, MS, and PD share multifaceted disabilities and underlying neuroinflammatory processes. The additional impact of COVID-19, especially in cases with persistent neurological manifestations, emphasizes the urgency of effective rehabilitation methods. Preliminary work by the research team includes studies on dual-task mechanisms and implementation in clinical settings, confirming feasibility and theoretical relevance. Nonetheless, rigorous randomized, controlled-possibly double-blind-trials are required to determine clinical efficacy.

Project Activities and Organization

The project includes the following integrated activities:

Design and validation of dual-task rehabilitation strategies, encompassing:

* dual motor tasks
* dual cognitive tasks
* combined motor-cognitive tasks Virtual and/or augmented reality environments will be used when beneficial. Pilot feasibility study in small groups (5 per diagnostic category: SO, MS, PD, long-term post-COVID) to assess applicability, patient acceptance, and preliminary efficacy. Conducted by OU1.

Participant selection for the clinical trial (SO, MS, PD, with or without past SARS-CoV-2 infection) based on predefined inclusion/exclusion criteria. Conducted jointly by all OUs.

Randomized controlled trial, conducted by OU1, OU3, and OU4, including:

1. Baseline motor, cognitive, and mood assessment using validated tools.
2. Implementation of dual-task strategies alongside standard rehabilitation, using emerging technological devices.
3. Re-assessment at treatment completion and at 3-month follow-up.

Data integration in a unified database (OU1). Statistical analyses and interpretation, including advanced methods such as artificial neural networks (OU1).

Dissemination through conferences and publications. Specific Aims Aim 1 - Development and feasibility testing of dual-task strategies

Dual-task interventions will be designed by OU1 based on the three task combinations. A preliminary feasibility phase will enroll 20 participants (5 SO, 5 MS, 5 PD, 5 post-COVID). Strategies demonstrating the best balance of efficacy and acceptability will be selected for the clinical trial.

Aim 2 - Application of validated strategies in a randomized controlled trial A total of 48 participants (16 SO, 16 MS, 16 PD) will be recruited; for each condition, half will have a history of SARS-CoV-2 infection with neurological symptoms persisting ≥4 weeks. Additional inclusion/exclusion criteria ensure safety and feasibility.

Participants will be randomized into:

* Experimental group: standard rehabilitation (3/week) with dual-task training (2/week, 30 min/session)
* Control group: standard rehabilitation with placebo low-resistance cycling (2/week, 30 min/session)

Aim 3 - Comparison of dual-task vs conventional rehabilitation outcomes

Outcome measures will be compared between:

* participants receiving standard with placebo therapy, and
* participants receiving standard with dual-task therapy.

Additionally, pre- and post-intervention blood samples will be analyzed for biomarkers of neuroinflammation and neurodegeneration, providing complementary insight into physiological changes associated with both rehabilitation modalities.

Appropriate statistical methods, including machine-learning-based analyses, will be used to evaluate between-group and within-group differences.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke outcomes, Multiple Sclerosis (MS), or Parkinson's disease (PD).
* For stroke outcomes: patients must be able to walk independently for at least 6 minutes without resting.
* For MS: diagnosis according to the 2017 revised McDonald criteria; relapsing-remitting or secondary progressive forms; age 25-65 years; Expanded Disability Status Scale score between 2.5 and 6.0.
* For PD: idiopathic Parkinson's disease.
* For each neurological condition, half of the participants must have had Severe Acute Respiratory Syndrome Coronavirus 2 infection with neurological symptoms attributable to CNS involvement lasting at least 4 weeks.
* Ability to provide informed consent.

Exclusion Criteria:

* Cognitive or motor comobidity;
* Severe visual or hearing impairments that may compromise understanding of exercises
* Language impairments, such as aphasia
* Inability to walk independently

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walking Test | Baseline (Day 1), end of treatment (Day 56), follow -up (146)
  The 6-Minute Walking Test is a standardized assessment of functional walking capacity in which the patient is instructed to walk back and forth along a predefined path for six minutes. The total distance covered during this time reflects the individual's aerobic endurance, mobility, and overall functional performance. The test is simple, well tolerated, and widely used in both clinical and research settings. The minimum score is about 300m and denotes a very low funcional motility, while higher distance covered (> 600 m) is a sign of good walking ability.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | Baseline (Day 1), End of Treatment (Day 56), 3-Month Follow-up (Day 146)
  The Montreal Cognitive Assessment is a widely used screening tool designed to evaluate global cognitive function. It assesses multiple domains, including attention, executive functions, memory, language, visuospatial abilities, abstraction, and orientation. The test is quick to administer, sensitive to mild cognitive impairment, and commonly applied in both clinical practice and research settings. The maximum score is 30, 25 is a cut off for normal cognitive functioning, with higher score denoting better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Iosa, PhD, Associate Professor, Principal Investigator — IRRCS Santa Lucia foundation
Locations (1):
- IRCCS Fondazione Santa Lucia, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No